CLINICAL TRIAL: NCT02843477
Title: Evaluation of Corrected Carotid Artery Flow Time as a Predictor of Fluid Responsiveness in Spontaneous Breathing Patients
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2016-0426
Record Dates: First submitted 2016-07-21; First posted 2016-07-25 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fluid loading group: Spontaneously breathing patients before induction of general anesthesia who receive fluid loading
  Interventions: Device: ultrasonographic measurement of corrected flow time in carotid artery

INTERVENTIONS:
Device: ultrasonographic measurement of corrected flow time in carotid artery — Corrected carotid artery flow time is measured using 10-5 MHz linear probe on a portable ultrasound machine. On the two-dimensional image, the optimal image of the long-axis view is obtained at the left common carotid artery. The sample volume is placed on the center of the lumen, 2 cm proximal to the bulb, and a pulsed wave Doppler examination was performed while the Doppler beams were adjusted to ensure < 60° of angle for the best signal. Then, cardiac cycle time and carotid flow time is measured. Carotid flow time is measured between the upstroke of the flow tracing and the dicrotic notch, and it is corrected for pulse rate by dividing flow time by the square root of the cardiac cycle time to calculate corrected carotid artery flow time (flow time/√cycle time).

SUMMARY:
It is still challenging to assess intravascular volume status in spontaneously breathing patients. Recently, the measurement of corrected flow time in carotid artery was introduced as quite useful, simple and noninvasive for the evaluation of circulating blood volume change. The aim of this study is to evaluate whether corrected carotid artery flow time as determined by ultrasonography can be a predictor of fluid responsiveness in spontaneously breathing patients before induction of general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (19-80 years of age) who were scheduled to undergo elective neurosurgery for brain tumor

Exclusion Criteria:

* BMI > 35 or < 15 kg/m2
* the presence of carotid artery stenosis > 50%
* systolic blood pressure > 160 mmHg
* cardiac rhythm other than sinus
* intracardiac shunt 6. valvular heart disease
* a left ventricular ejection fraction of < 50%
* right ventricular dysfunction 9
* chronic obstructive pulmonary disease
* pulmonary hypertension
* chronic kidney disease (eGFR < 60 mL/min/1.73m2)
* pregnancy

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were scheduled to undergo elective neurosurgery for brain tumor
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2016-08-09 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
ultrasonographic measurement of corrected flow time in carotid artery | right before fluid loading
  The ultrasonographic measurement of corrected flow time in carotid artery will be performed before fluid loading.
ultrasonographic measurement of corrected flow time in carotid artery | 5 minutes after fluid loading
  The ultrasonographic measurement of corrected flow time in carotid artery will be performed 5 minutes after fluid loading.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim DH, Shin S, Kim N, Choi T, Choi SH, Choi YS. Carotid ultrasound measurements for assessing fluid responsiveness in spontaneously breathing patients: corrected flow time and respirophasic variation in blood flow peak velocity. Br J Anaesth. 2018 Sep;121(3):541-549. doi: 10.1016/j.bja.2017.12.047. Epub 2018 Apr 12. PMID 30115251